CLINICAL TRIAL: NCT06977386
Title: The Application Value of Spectral CT in the Accurate Staging of Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLX2025-102
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The application value of spectral CT in the accurate staging of gastric cancer (Experimental): Prospectively collect medical images and clinical data related to gastric cancer using Philips Quark CT equipment, and evaluate the diagnostic accuracy and clinical application value in the accurate staging of gastric cancer.Patients diagnosed with gastric cancer in Yunnan Provincial Cancer Hospital from April 2025 to May 2026 were consecutively included, and after scanning with Philips Quark CT, the TNM stage of gastric cancer patients was assessed by two radiologists, and finally statistical analysis was performed.
  Interventions: Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of gastric cancer

INTERVENTIONS:
Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of gastric cancer — CT scan of the abdomen outside of standard treatment options

SUMMARY:
Spectral CT was used to prospectively collect medical images and clinical data related to gastric cancer, evaluate the effect of image quality in the diagnosis of gastric cancer, and evaluate the application value in the accurate staging of gastric cancer, so as to provide a more accurate clinical basis for diagnosis, promote the development of individualized treatment, and ultimately improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* (a)Patients with pathologically confirmed gastric cancer;
* (b) aged ≥ 18 years old;
* (c) have not received chemoradiotherapy or surgery.

Exclusion Criteria:

* (a)Combined with other primary tumors;
* (b) The image quality does not meet the diagnostic criteria;
* (c)Those who cannot tolerate CT examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological TNM staging | 1 day
  Pathological examination information: The pathology results using surgery/biopsy data are the gold standard, and the depth of tumor invasion, lymph node metastasis, and distant metastasis are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China